CLINICAL TRIAL: NCT06466863
Title: Cultural Adaptation, Validity, and Reliability Study of the Turkish Version of the Youth Activity Profile (YAP-Turkey)
Brief Title: Turkish Cultural Adaptation, Validity and Reliability Study of Youth Activity Profile
Acronym: YAP-Turkey
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Asst.prof, Istanbul University - Cerrahpasa
Other Study IDs: 67G2qhEM
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Physical Activity; Children
Keywords: physical activity; children; Yap; Turkish Version
MeSH Terms: conditions — Motor Activity | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Our study will be conducted as a single-group design: This study will be conducted with healthy young people aged 12-17 years who voluntarily agree to participate in the study. Individuals will be included in the study after obtaining consent from the participants and their parents.
  This questionnaire will be filled in at the convenience of the participants during the academic year. Then the questions of the Youth Activity Profile (YAP) will be asked. The time required to complete the questionnaires is approximately 20 minutes in total.
  Interventions: Other: Validity and Reliability

INTERVENTIONS:
Other: Validity and Reliability — Participants were included in the study after obtaining consent from both the participants and their parents. Participants were informed about the study prior to the survey, and only those who volunteered were included in the study. The data collection process was conducted online via Google Forms. The assessment form was sent to the participants through social media platforms, messages, and emails. Participants completed the YAP-T twice, 7 days apart, and all measurements were taken on weekdays under similar conditions by the same evaluators (4 evaluators) in the same region (Istanbul).
  Test-retest reliability will be determined by calculating the Intraclass Correlation Coefficient (ICC) between the total scores obtained from the two assessments.

SUMMARY:
Aim: The aim of this study is to conduct a Turkish cultural adaptation, validity, and reliability study of the Youth Activity Profile (YAP), developed to assess physical activity and sedentary behavior in a sample of individuals aged 12-17 years of Turkish descent.

Method: Online surveys will be distributed to participants through social media platforms, messages, and emails. Participants' demographic information will be obtained using an online assessment form prepared by the researchers. Subsequently, the Physical Activity Questionnaire for Adolescents (PAQ-A) will be used to determine the levels of physical activity. This survey will be completed by participants at a time convenient for them during the academic term. Following this, questions from the Youth Activity Profile (YAP) will be administered. Once the targeted number of participants is reached, the data collection process will be concluded, and the survey link will be deactivated.

Potential Outcomes: It is expected that this study will contribute to a better understanding of the health behaviors and physical activity trends of adolescents aged 12-17 years, thereby informing health policies.

DETAILED DESCRIPTION:
Adolescence represents a critical developmental period during which individual lifestyle preferences and behavioral patterns are formed. According to the World Health Organization (WHO), the age range of 10-19 years is defined as the adolescent period. Regular physical activity (PA) is crucial for maintaining health during this period. WHO recommends that children and adolescents aged 5-17 years engage in moderate to high-intensity physical activity for at least 60 minutes a day. However, it is reported that globally, 80.3% of adolescents do not reach the recommended PA level. Studies have indicated an increase in the prevalence of diseases such as obesity, mental health problems, and hypertension during adolescence, highlighting the critical importance of physical activity during this phase. Therefore, accurate assessment of PA and sedentary behavior (SB) is essential. Self-report questionnaires, as subjective methods, provide an accurate and reliable means to define the PA/SB ratio and also offer a more cost-effective evaluation opportunity. It is believed that evaluating personal factors such as gender, age, and weight, along with contextual factors both in and out of school, is important in assessing the physical activity level and quality of adolescents.

Currently, there is no specific questionnaire validated and reliable in Turkish that covers the age range of 12-17 years for assessing PA and SB levels. Studies have shown that the methodological quality and validity of commonly used questionnaires to measure PA and SB in adolescents have some limitations. Therefore, further research is necessary to enhance and standardize surveys in this field in Turkey. These studies are crucial for better understanding the health behaviors and trends among young people and for guiding health policies.

The aim of this study was to conduct a Turkish cultural adaptation, validity, and reliability study of the Youth Activity Profile (YAP), developed to assess physical activity and sedentary behavior in adolescents within a sample of Turkish individuals aged 12-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 17
* Enrolled in primary or middle school
* Volunteering to participate in the study

Exclusion Criteria:

* Having any serious visual impairment or mental health problem
* Not having the ability to read and write in Turkish
* Having any orthopedic, neurological, or rheumatological disease that may affect physical activity levels

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged between 12 and 17, both male and female, attending primary or middle school.
  In order to determine the validity and reliability of the scale, the number of items of the tested scale was taken into consideration in determining the sample number to be included in the study (15 items in total). The number of volunteers was determined as ten times the number of items (150 participants) and 15 substitutes were added to the number of volunteers considering the drops and the number of the sample was determined as 165.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Youth Activity Profile (YAP) | Change from baseline to 7 day
  The Youth Activity Profile (YAP) is a 15-item questionnaire developed to evaluate physical activity and sedentary behavior in children and adolescents aged 8 to 17 years. It operates on a recall basis, covering activities over the previous week (7 days) and includes assessments of both school and out-of-school activities, as well as time spent in sedentary behaviors.

SECONDARY OUTCOMES:
Physical Activity Questionnaire for Adolescents (PAQ-A) | Baseline
  The scale consisting of 10 questions is calculated with a 5-point Likert system. The 1st question is divided into 15 items. In the calculation of the 1st question, the result obtained by dividing each score given for 15 items by the number of items is used. The scores given for each of the questions 2-8 are totalled. The 9th question consists of 7 items in total

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman Arman, Asst. Prof., Principal Investigator — Istanbul University-Cerrahpasa Istanbul, Turkey

IPD SHARING:
Plan to Share IPD: Undecided